CLINICAL TRIAL: NCT01423643
Title: HCV/HIV Coinfection: Antiviral Therapy and Fibrosis
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Thomas, Chief, Infectious Diseases, Johns Hopkins University
Other Study IDs: NA00033421; R01DA013806 (NIH)
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infection; Hepatitis C
Keywords: HIV; Human immunodeficiency virus; Acquired Immune Deficiency Syndrome Virus; AIDS Virus; Immunodeficiency Virus, Human; Virus, Human Immunodeficiency; Hepatitis C; Hepatitis C, chronic; Hepatitis C virus; Hepatitis C antibodies; Hepatitis C antigens
MeSH Terms: conditions — HIV Infections; Hepatitis C; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen serum and plasma samples. Liver biopsy fixed slides.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Main cohort: Adults infected with both HIV and Hepatitis C
- Control Group: Adults at risk for liver disease, but not infected with both HIV and Hepatitis C

SUMMARY:
The chief purpose of this research is to understand how antiretroviral therapy (ART) affects progression of liver disease in persons co-infected with HIV and hepatitis C virus (HCV). The investigators study liver disease progression in a cohort of dually infected persons according to the success of ART.

DETAILED DESCRIPTION:
Enrolled subjects will complete questionnaires concerning health status, lifestyle, and alcohol/drug use. Participants will undergo liver elastography every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

Co-Infected Arm

1. Subject must be an HIV/HCV co-infected adult with HIV infection diagnosed by antibody testing and chronic HCV infection diagnosed by reactive HCV antibody and detectable plasma HCV RNA.
2. Subject must receive medical care at the JHU HIV clinic or through the Viral Hepatitis Center.
3. Subjects previously enrolled in the study cohort, but not currently receiving care in the Moore Clinic, may continue in the study.
4. Females of childbearing potential must be willing to undergo a urine or serum pregnancy test.
5. Subject must be able to provide informed written consent.

Control Arm

1. Subject must have or be at risk of having medical conditions that increase the risk of liver disease. These include, but are not limited to, HIV mono-infection, HCV mono-infection, Hepatitis B infection, alcohol addiction, and/or non-alcoholic steatohepatitis.
2. Females of childbearing potential must be willing to undergo a urine or serum pregnancy test.
3. Subject must be able to provide informed written consent.

Exclusion Criteria:

1. To avoid risks associated with ionizing radiation, female subjects may not be pregnant or breast feeding at the time of DEXA scanning. To avoid unknown risks to the fetus, female subjects may not be pregnant at the time of liver biopsy or FibroScan.
2. To avoid interference with the DEXA scan, the subject may not have undergone a nuclear medicine exam with the past week and/or may not have undergone an x-ray procedure with contrast solution within the past 72 hours.
3. To avoid unknown risks, subjects with an implanted cardiac device such as a defibrillator or pacemaker may not undergo FibroScan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with HIV and Hepatitis C in the metropolitan Baltimore area. Preference given to those enrolled in the Johns Hopkins Infectious Diseases Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2001-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Fibrosis stage | up to 15 years
  Liver histologic fibrosis stage (Ishak 0 - 6)

SECONDARY OUTCOMES:
Body composition | up to 15 years
  Body composition measurements, derived from DEXA
Liver stiffness | up to 15 years
  Liver stiffness, derived from liver elastography
Serum markers | up to 15 years
  Serum levels of various chemical markers
Liver histology | up to 15 years
  Liver histology as described by a pathologist

CONTACTS AND LOCATIONS:
Overall Officials: David L. Thomas, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Salgado M, Kirk GD, Cox A, Rutebemberwa A, Higgins Y, Astemborski J, Thomas DL, Thio CL, Sulkowski MS, Blankson JN. Protective interleukin-28B genotype affects hepatitis C virus clearance, but does not contribute to HIV-1 control in a cohort of African-American elite controllers/suppressors. AIDS. 2011 Jan 28;25(3):385-7. doi: 10.1097/QAD.0b013e328341b86a. PMID 21099664
- [Background] Brown TT, Mehta SH, Sutcliffe C, Higgins Y, Torbenson MS, Moore RD, Thomas DL, Sulkowski MS. Hepatic steatosis associated with increased central body fat by dual-energy X-ray absorptiometry and uncontrolled HIV in HIV/hepatitis C co-infected persons. AIDS. 2010 Mar 27;24(6):811-7. doi: 10.1097/QAD.0b013e3283333651. PMID 20186036
- [Background] Balagopal A, Ray SC, De Oca RM, Sutcliffe CG, Vivekanandan P, Higgins Y, Mehta SH, Moore RD, Sulkowski MS, Thomas DL, Torbenson MS. Kupffer cells are depleted with HIV immunodeficiency and partially recovered with antiretroviral immune reconstitution. AIDS. 2009 Nov 27;23(18):2397-404. doi: 10.1097/QAD.0b013e3283324344. PMID 19773633
- [Background] Kirk GD, Astemborski J, Mehta SH, Spoler C, Fisher C, Allen D, Higgins Y, Moore RD, Afdhal N, Torbenson M, Sulkowski M, Thomas DL. Assessment of liver fibrosis by transient elastography in persons with hepatitis C virus infection or HIV-hepatitis C virus coinfection. Clin Infect Dis. 2009 Apr 1;48(7):963-72. doi: 10.1086/597350. PMID 19236273
- [Result] El-Maouche D, Mehta SH, Sutcliffe C, Higgins Y, Torbenson MS, Moore RD, Thomas DL, Sulkowski MS, Brown TT. Controlled HIV viral replication, not liver disease severity associated with low bone mineral density in HIV/HCV co-infection. J Hepatol. 2011 Oct;55(4):770-6. doi: 10.1016/j.jhep.2011.01.035. Epub 2011 Feb 19. PMID 21338640
- [Result] Woreta TA, Sutcliffe CG, Mehta SH, Brown TT, Higgins Y, Thomas DL, Torbenson MS, Moore RD, Sulkowski MS. Incidence and risk factors for steatosis progression in adults coinfected with HIV and hepatitis C virus. Gastroenterology. 2011 Mar;140(3):809-17. doi: 10.1053/j.gastro.2010.11.052. Epub 2010 Dec 4. PMID 21134375
- [Result] Sulkowski MS, Mehta SH, Torbenson MS, Higgins Y, Brinkley SC, de Oca RM, Moore RD, Afdhal NH, Thomas DL. Rapid fibrosis progression among HIV/hepatitis C virus-co-infected adults. AIDS. 2007 Oct 18;21(16):2209-16. doi: 10.1097/QAD.0b013e3282f10de9. PMID 18090048
- [Result] Mehta SH, Lucas GM, Mirel LB, Torbenson M, Higgins Y, Moore RD, Thomas DL, Sulkowski MS. Limited effectiveness of antiviral treatment for hepatitis C in an urban HIV clinic. AIDS. 2006 Nov 28;20(18):2361-9. doi: 10.1097/QAD.0b013e32801086da. PMID 17117023